CLINICAL TRIAL: NCT03866525
Title: Phase I/II Study of OH2 Injection, an Oncolytic Type 2 Herpes Simplex Virus Expressing Granulocyte Macrophage Colony-Stimulating Factor, in Malignant Solid Tumors
Brief Title: OH2 Oncolytic Viral Therapy in Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Binhui Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OH2-I-ST-02
Record Dates: First submitted 2019-02-28; First posted 2019-03-07 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumor; Gastrointestinal Cancer
Keywords: Oncolytic Virus
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose escalation and dose expansion (Experimental): A 3+3 dose-escalation strategy is used in the phase 1 part and 3 dose levels (10e6, 10e7 and 10e8 CCID50/mL) of OH2 are assessed as single agent and in combination with HX008. The recommended dose levels are then determined and adopted in the phase 2 part for dose-expansion.
  In the phase 2 dose-expansion part, OH2 will be delivered as single agent in cohort 1, in combination with irinotecan in cohort 2, in combination with HX008 in cohort 3 and 4. There are no comparator arms for these cohorts.
  Interventions: Biological: OH2 injection, with or without irinotecan or HX008

INTERVENTIONS:
Biological: OH2 injection, with or without irinotecan or HX008 — OH2: Oncolytic Type 2 Herpes Simplex Virus Irinotecan: cytotoxic agent HX008: anti-PD-1 antibody

SUMMARY:
This phase I/II study evaluates the safety and efficacy of OH2 as single agent or in combination with HX008, an anti-PD-1 antibody, in patients with malignant solid tumors (gastrointestinal cancers, head and neck cancers, soft tissue sarcomas).

OH2 is an oncolytic virus developed upon genetic modifications of the herpes simplex virus type 2 strain HG52, allowing the virus to selectively replicate in tumors. Meanwhile, the delivery of the gene encoding human granulocyte macrophage colony-stimulating factor (GM-CSF) may induce a more potent antitumor immune response.

DETAILED DESCRIPTION:
This is a phase I/II study evaluating the safety and efficacy of OH2 injection in patients with malignant solid tumors.

In the phase I dose escalation part, three doses (1x10e6, 1x10e7, 1x10e8 CCID50/mL) of OH2 will be delivered intratumorally as single agent and in combination with HX008 to observe the DLTs and to identify the MTD. After the completion of phase I, the recommended dose for single agent and combination therapy will be determined for dose expansion in phase II.

The phase II part comprises of 4 cohorts. In cohort 1, patients will be treated at the recommended dose as defined in phase 1. In cohort 2, OH2 will be delivered in combination with irinotecan for the treatment of advanced gastrointestinal cancers. In cohort 3, OH2 will be injected in combination with HX008, and the first doses of the two anti-tumor agents will be administered on the same day. The treatments in cohort 4 will be identical as in cohort 3, except that the first dose of HX008 will be administered at the time of the third dose of OH2.

The biodistribution of OH2 is evaluated in the phase 1 part of the trial by detection of viral loads in the blood, urine, and saliva at different timepoints. In addition, the injection sites are swabbed for virus shedding on the next day of each dose from cycle 1-3.

Adverse events (AEs) and DLTs are graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0). Radiographic imaging studies are performed using computed tomography or magnetic resonance imaging. Measurement of cutaneous or subcutaneous lesions are conducted with calipers. Evaluation of response are performed by the investigators using both the RECIST version 1.1 and the iRECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed unresectable or recurrent/metastatic solid tumors.
2. The patient must have failed the standard treatment (due to either disease progression or intolerable toxicity) or the standard of care had not been established for the specific condition.
3. Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
4. Eastern Collaborative Oncology Group (ECOG) Performance Status ≤ 1.
5. Life expectancy >3 months.
6. The patient must have at least one tumor site appropriate for intratumoral injection.
7. Adequate organ function.
8. Participants of reproductive potential must be willing to use adequate contraception for the course of the study until 3 months after the last dose of any of the drugs in the study.
9. Participants with a history of HSV infection must have recovered at least 3 months before the study.
10. Willing and able to provide written informed consent and comply with the requirements of the study.

Exclusion Criteria:

1. Uncontrolled concurrent illness including, but not limited to, severe cardiac disease, cerebralvascular disease, uncontrolled diabetes, uncontrolled hypertension, ongoing or active systemic infection, active peptic ulcer disease.
2. Central nervous system (CNS) metastases with clinical symptoms
3. Active infection or an unexplained fever > 38.5°C.
4. Known Human Immunodeficiency Virus (HIV) infection, active Hepatitis B or Hepatitis C infection.
5. Pregnant or lactating female.
6. Patients who are receiving any other investigational agents.
7. Known immediate or delayed hypersensitivity reaction to HSV.
8. Previous malignancy within 5 years prior to study entry.
9. Patients with any active autoimmune disease or history of autoimmune disease.
10. Concurrent medical condition requiring the use of cortisol (>10mg/day prednisone or equivalent dose) or other systematic immunosuppressive medications within 14 days before the study treatment, except for inhalation or topical corticosteroids no more than 10 mg/day prednisone or equivalent.
11. Familial, sociological or geographical conditions that, in the judgment of the investigator, do not permit compliance with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
The dose-limiting toxicities (DLTs) of OH2 injection as single agent and in combination with HX008 in patients with solid tumors | 6 months
  Primary outcome of phase 1.
The maximum-tolerated doses (MTDs) of OH2 injection as single agent and in combination with HX008 in patients with solid tumors | 6 months
  Primary outcome of phase 1.
The biodistribution and biologic effect of OH2 injection | 6 months
  Primary outcome of phase 1. The biodistribution of OH2 is evaluated by detection of viral loads in the blood, urine, and saliva. Additionally, the injection sites are swabbed for virus shedding. For the analyses of biologic effects, serum samples are collected for HSV serology assays and assessment of GM-CSF protein and GM-CSF RNA.
The anti-tumor activity of OH2 monotherapy and in combination with irinotecan or HX008 | 2 years
  Primary outcome of phase 2.

SECONDARY OUTCOMES:
The anti-tumor activity of OH2 monotherapy and in combination with HX008 | 2 years
  Secondary outcome of phase 1.
The immunogenicity of OH2 | 2 years
  Secondary outcome of phase 1. The immunogenicity of OH2 is evaluated by detection of anti-GM-CSF antibodies in the blood.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request are accessible from Binhui Biotech. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in China or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement.

REFERENCES:
- [Derived] Wang Y, Jin J, Li Y, Zhou Q, Yao R, Wu Z, Hu H, Fang Z, Dong S, Cai Q, Hu S, Liu B. NK cell tumor therapy modulated by UV-inactivated oncolytic herpes simplex virus type 2 and checkpoint inhibitors. Transl Res. 2022 Feb;240:64-86. doi: 10.1016/j.trsl.2021.10.006. Epub 2021 Oct 29. PMID 34757194